CLINICAL TRIAL: NCT05003479
Title: A Randomized, Double-blind, Placebo-controlled Phase Ⅰ Clinical Study to Evaluate the Safety and Immunogenicity of SARS-CoV-2 Vaccine (Vero Cells), Inactivated in Healthy Population Aged 3 to 17 Years
Brief Title: Clinical Trial of SARS-CoV-2 Vaccine (Vero Cells), Inactivated in Healthy Population Aged 3 to 17 Years(COVID-19)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Kangtai Biological Products Co., LTD (Industry)
Collaborators: Beijing Minhai Biotechnology Co., Ltd (Industry); Hunan Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020L001-2A
Record Dates: First submitted 2021-08-10; First posted 2021-08-12 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- candidate vaccine (Experimental)
  Interventions: Biological: SARS-CoV-2 Vaccine (Vero Cells), Inactivated
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SARS-CoV-2 Vaccine (Vero Cells), Inactivated — 2 doses of SARS-CoV-2 Vaccine (Vero Cells), Inactivated should be administered as an intramuscular injection into the lateral deltoid of the upper arm with a 28-day interval.
  Arms: candidate vaccine
Biological: Placebo — 2 doses of Placebo should be administered as an intramuscular injection into the lateral deltoid of the upper arm with a 28-day interval.
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blinded, and placebo controlled phase Ⅰ clinical trial of the SARS-CoV-2 inactivated vaccine to evaluate the safety and immunogenicity of the experimental vaccine in healthy population aged 3 to 17 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy residents aged 3 to 17 years at the time of consent
* Subjects and/or their guardian agree to sign the informed consent forms voluntarily.
* Be able to comply with study requirements/procedures.
* Axillary temperature ≤ 37.0℃

Exclusion Criteria:

* Within 14 days before vaccination, subjects have been abroad and to villages/communities experienced COVID-19 epidemics, and in contact with COVID-19 cases or suspected cases. Subjects are under isolation observation, or living in the villages/communities with COVID-19 cases or suspected cases;
* Confirmed cases, suspected cases or asymptomatic cases with COVID-19 (refer to Information System of China Disease Prevention and Control);
* Subjects with history of SARS virus infection by self-reported;
* Positive in throat swab through RT-PCR;
* History of vaccination of various COVID-19 vaccines or positive in SARS-CoV-2 antibody test;
* Positive urine pregnancy test for females with menarche
* With abnormal indicators, such as blood biochemistry, blood routine, urine routine, thyroid function and coagulation function which might show clinical meaning, before administration;
* History of severe allergic reactions (such as acute anaphylaxis, urticaria, skin eczema, dyspnea, angioneurotic edema or abdominal pain) or allergy to known composition of inactivated SARS-CoV-2 vaccine;
* History or family history of convulsion, epilepsy, encephalopathy or mental illness;
* Subjects with congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Subjects with known or suspected diseases include: severe respiratory diseases, severe cardiovascular diseases, severe liver and kidney diseases, drug-uncontrollable hypertension, diabetic complications, malignant tumors, various acute diseases or acute onset of chronic diseases;
* Diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases;
* History of coagulation dysfunction (e.g. Coagulation factor deficiency, coagulation disease);
* Subjects receiving anti-TB treatment;
* Subjects receiving other research drugs within 6 months before vaccination;
* Subjects receiving immunotherapy or inhibitor therapy within 3 months (consistently oral or infusion for more than 14 days);
* Subjects receiving blood products within 3 months before administration;
* Subjects vaccinated with live attenuated vaccine within 14 days before vaccination;
* Subjects vaccinated with other vaccine within 7 days before vaccination;
* The researchers shall judge the other conditions which might be not in compliance with the requirements of this clinical trial.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse reactions/events | 0-28 days after each vaccination

SECONDARY OUTCOMES:
Incidence of Serious Adverse Events (SAE) | within 12 months post full vaccination
Incidence of abnormal indicators of laboratory safety examinations(including blood routine, blood biochemistry, urine routine, thyroid function and coagulation function) | Day 3 after each dose of vaccination
Geometric mean titer of SARS-CoV-2 neutralizing antibody | 28 days, 3 months, 6 months and 12 months post full vaccination
Geometric mean titer of SARS-CoV-2 IgG binding antibody | 28 days, 3 months, 6 months and 12 months post full vaccination
Seroconversion rate of SARS-CoV-2 neutralizing antibody | 28 days post full vaccination
Seroconversion rate of SARS-CoV-2 IgG binding antibody | 28 days post full vaccination
Seropositive rate of SARS-CoV-2 neutralizing antibody | 3 months, 6 months and 12 months post full vaccination
Seropositive rate of SARS-CoV-2 IgG binding antibody | 3 months, 6 months and 12 months post full vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial Center for Diseases Control and Prevention, Changsha, Hunan, China

REFERENCES:
- [Derived] Liu J, Huang B, Li G, Huang T, Wang D, Zhang L, Deng Y, Chang X, Liu Y, Li W, Zhang S, Huang W, Tan W, Gao L. Immunogenicity and Safety of a SARS-CoV-2 Inactivated Vaccine KCONVAC in Chinese Children: Randomized, Double-blind, Placebo-controlled Phase 1 and 2 Trials. Pediatr Infect Dis J. 2023 Dec 1;42(12):1136-1142. doi: 10.1097/INF.0000000000004085. Epub 2023 Sep 4. PMID 37967148